CLINICAL TRIAL: NCT05448118
Title: Virtual MOUD Treatment: Virtual Point-of-Care Toxicology Testing to Accompany Virtual Medication Assisted Treatment for Opioid Use Disorder
Brief Title: Virtual MOUD Treatment- Virtual POC Toxicology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This Pilot implementation Trial was never started because no providers were found who would agree to use saliva-based toxicology tests in care
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SDR 21-114
Record Dates: First submitted 2022-06-24; First posted 2022-07-07 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Substance Use Disorder
Keywords: Substance Use Disorder; Opioid Use Disorder; Telemedicine; Toxicology
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: A virtual point-of-care toxicology testing process will be evaluated in a single arm pilot trial among providers and patients at VACT and VACWM. Acceptability will be evaluated through patient and provider semi-structured interviews. Overall feasibility will be determined by evaluating virtual toxicology testing utilization, as well as the frequency of toxicology testing and of addiction treatment contacts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual POC Toxicology Testing (Experimental): Providers and patients will use Saliva Toxicology test at the point of care during virtual care visits.
  Interventions: Diagnostic Test: Virtual POC Toxicology Test

INTERVENTIONS:
Diagnostic Test: Virtual POC Toxicology Test — Providers and patients will use Saliva Toxicology test at the point of care during virtual care visits.

SUMMARY:
Care for Substance use disorders (SUD) such as Medication treatment of Opioid Use Disorder (MOUD) saves lives and is increasingly delivered virtually. Currently, 60% of VA outpatient addiction treatment occurs over video. However, toxicology testing, a major component of SUD care, currently requires in-person visits. A process for virtual point-of-care toxicology testing is needed. This research will develop a Virtual Point-of-Care Toxicology Testing Process for VA. This Pilot Trial will evaluate the feasibility, acceptability, and proximal effects of the process by evaluating provider and patient testing uptake, qualitative feedback, and health service use.

DETAILED DESCRIPTION:
Care for Substance use disorders (SUD) such as Medication treatment of Opioid Use Disorder (MOUD) saves lives and is increasingly delivered virtually. Currently, 60% of VA outpatient addiction treatment occurs over video. However, toxicology testing, a major component of MOUD care, currently requires in-person visits. A process for virtual point-of-care toxicology testing is needed. The objectives of this pilot project are to develop, feasibility test, and describe the proximal outcomes of a Virtual Point-of-Care Toxicology Testing Process for VA patients in MOUD care.

The process will be evaluated in a pilot trial among providers and patients at VA Connecticut (VACT) and VA Central Western Massachusetts (VACWM). Acceptability will be evaluated through patient and provider semi-structured interviews. Overall feasibility will be determined using a priori benchmarks of utilization. These findings will be used to inform modifications of virtual toxicology testing procedures.

Mixed-methods will be used to develop and evaluate the testing process, which will use an oral-fluid test for common drugs of abuse. The test is FDA approved for at home patient use. Patients will self-administer the test during virtual SUD visits and assess results with providers. In the pilot trial, a single-arm mixed-methods pilot trial will evaluate the process among patients and providers at two VA facilities. Feasibility will be evaluated by examining process uptake. Acceptability will be evaluated through semi-structured interviews with patients and providers based on Consolidated Framework for Implementation Research (CFIR) constructs. Health service use will be evaluated by analyzing data on patient characteristics, test utilization, and treatment contacts extracted from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

To participate VA patients must

* be recruited by their provider through a discussion about the project
* be interested in participating after the discussion
* have used VA video-based care at least once
* receive buprenorphine from a VACT or VAWCM provider (50% will have started buprenorphine within the last 3 months)
* have the ability to receive mail from the VA for the purposes of receiving oral fluid test kits)

Exclusion Criteria:

* Veterans must not be receiving inpatient or day-program treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure | at enrollment and between 2 and 3 months following enrollment
  The Acceptability of intervention measure is a 4-item measure scored on a 5-point scale and summed. The Range of Scores is from 4 to 20. Higher Scores indicate higher acceptability.
Semi-Structured Interview of Toxicology Testing Process Acceptability | Through study completion or 3-months post enrollment, whatever comes first
  Semi-Structured interview of toxicology testing Process Acceptability based on the Consolidated Framework for Implementation Research, transcribed and analyzed qualitatively for key themes.

SECONDARY OUTCOMES:
The Substance Abuse Perceived Stigma Scale | at enrollment and between 2 and 3 months following enrollment
  The Substance Abuse Perceived Stigma Scale (SAPSS) is a 12-item questionnaire that assesses the construct of perceived stigma. Items are scored on seven point Likert-type scale where 1 = never and 7 = always with agreement indicating non-stigmatizing behavior or attitudes. The scale is scored by reverse scoring each item, summing the items, and dividing by 12, thus higher scores indicate more perceived stigma.
Helping Alliance questionnaire | at enrollment and between 2 and 3 months following enrollment
  Helping Alliance questionnaire (HAq-II) is a 19-item questionnaire that measures the strength of the patient-therapist therapeutic alliance. Each item is rated on a 6-point Likert scale (1 = I strongly feel it is not true, 6 = I strongly feel it is true). Negatively worded items are reverse scored.
Health service use | 6 months following enrollment
  toxicology testing episodes and substance use disorder treatment contacts will be extracted from the electronic medical record. Toxicology testing episodes will be measured as a proportion of SUD treatment encounters over a 6 month period following enrollment and Substance use disorder treatment contacts will be summed over a 6 month period following enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hermes, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts

IPD SHARING:
Plan to Share IPD: No